CLINICAL TRIAL: NCT00034723
Title: MRI Investigation Of The CNS In HTLV-1 Associated Myelopathy/Tropical Spastic Paraparesis (HAM/TSP)
Brief Title: MRI Brain Studies in Patients With HTLV-1 Associated Myelopathy/Tropical Spastic Paraparesis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020180; 02-N-0180
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-03

CONDITIONS: Tropical Spastic Paraparesis
Keywords: DTI; MRSI; MTR; NAWN; Fiber-Tract; Normal Control; Healthy Volunteer; HV; HTLV-1 Associated Myelopathy; Tropical Spastic Paraparesis; HAM/TSP
MeSH Terms: conditions — Paraparesis, Tropical Spastic

SUMMARY:
This study will use three different magnetic resonance imaging (MRI) techniques to study HTLV-1 associated myelopathy/tropical spastic paraparesis (HAM/STP)-a disease of slowly progressive weakness in the legs. It is not known how the HTLV-1 virus causes this disease, but it is thought that as the body's immune system tries to destroy the virus, parts of the nervous system-primarily the spinal cord-are damaged.

Patients 18 years of age and older with HAM/TSP and healthy normal volunteers may be eligible for this study.

Participants will undergo diffusion tensor MRI, MR-spectroscopy, and magnetization transfer imaging to look at different compositional, architectural, and microscopic properties of the brain. All of these techniques are similar to conventional MRI, and like the conventional method they use a strong magnetic field and radio waves to measure structural and chemical changes in brain tissue. Each of the three scans will be done on separate days, each lasting about 1 hour. For the procedures, the patient or volunteer lies on a stretcher in a narrow metal cylinder (the scanner) and is asked to remain still for 15 to 30 minutes at a time. A special lightweight coil may be placed on the head to enhance the brain images. The subject can communicate with the person doing the scan at all times.

DETAILED DESCRIPTION:
Magnetic Resonance Imaging (MRI) has become an important tool in the diagnosis of inflammatory CNS diseases such as Multiple Sclerosis (MS) and HTLV-1 Associated Myelopathy/Tropical Spastic Paraparesis (HAM-TSP). It is widely used as a marker for disease activity and progression. However, conventional MRI methods are only suitable to study gross anatomical features, such as size and shape of a particular area of the brain; questions regarding intrinsic microstructure and morphologic specificity cannot be addressed. But axonal damage or structural abnormalities even in normal appearing brain tissue may play an important role in the development of irreversible disability. Magnetization Transfer Imaging, Magnetic Resonance Spectroscopy and Diffusion Tensor MRI are imaging techniques described to be capable of the detection of such changes. Spectroscopy can detect molecular components in tissue, whereas the Magnetization Transfer Ratio (MTR) allows the measurement of water-macromolecule interactions. Diffusion Tensor MRI (DT-MRI) is an imaging modality that combines features of in vivo anatomical MRI and histopathology: it is an in vivo MRI method that provides information about tissue composition, microstructure, organization and architecture. This is possible because water diffusion properties in tissues, as measured by DT-MRI, are affected by tissue constituents, such as macromolecules, membranes, organelles, as well as by tissue microstructure, architecture and organization. A study comprising Magnetization Transfer-, Spectroscopy- and DT-MRI furnishes important information that cannot be obtained using conventional MRI methods.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients:

A. Established Diagnosis of HAM/TSP as defined by Osame, Igata, and Matsumoto and subsequently confirmed by Gessain and Gout and the WHO.

B. Age 18 or older

C. An initial cohort of 5 HAM/TSP patients with established disease with EDSS levels of 6.0 or greater and duration of disease of 2 years or more will be investigated. If MRI abnormalities can be demonstrated, the group will be expanded to 20. Of this 20, at least 5 patients have been identified that will be HLA A201.

Healthy Controls:

A. No history of disease of the nervous system or autoimmune disease

B. Age 18 or older

C. Subjects shall be sex- and age-matched to our patients

EXCLUSION CRITERIA:

A subject will be excluded if he/she has a contraindication to MRI scanning such as the following: Aneurysm clip; Implanted neural stimulator; Implanted cardiac pacemaker or autodefibrillator; Cochlear implant; Ocular foreign body or implant (e.g. metal savings, retinal clips); breast implants; or Insulin pumps. Subjects will be excluded if they have claustrophobia. A pregnancy test will be administered to women of childbearing age. Pregnant women will be excluded from the studies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2002-04; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] McDonald WI, Compston A, Edan G, Goodkin D, Hartung HP, Lublin FD, McFarland HF, Paty DW, Polman CH, Reingold SC, Sandberg-Wollheim M, Sibley W, Thompson A, van den Noort S, Weinshenker BY, Wolinsky JS. Recommended diagnostic criteria for multiple sclerosis: guidelines from the International Panel on the diagnosis of multiple sclerosis. Ann Neurol. 2001 Jul;50(1):121-7. doi: 10.1002/ana.1032. PMID 11456302
- [Background] Frank JA, McFarland HF. How to participate in a multiple sclerosis clinical trial. Neuroimaging Clin N Am. 2000 Nov;10(4):817-30 ,x. PMID 11359727
- [Background] Gessain A, Gout O. Chronic myelopathy associated with human T-lymphotropic virus type I (HTLV-I). Ann Intern Med. 1992 Dec 1;117(11):933-46. doi: 10.7326/0003-4819-117-11-933. PMID 1443956